CLINICAL TRIAL: NCT02060032
Title: COMPARATIVE EVALUATION OF CLINICAL EFFICACY OF SUBGINGIVALLY DELIVERED 1.2% ATORVASTATIN AND 1.2% SIMVASTATIN IN TREATMENT OF CHRONIC PERIODONTITIS: A RANDOMIZED CONTROLLED TRIAL
Brief Title: 1.2% Atorvastatin and 1.2% Simvastatin in Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2011-2012/B
Record Dates: First submitted 2014-02-05; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Periodontitis
Keywords: Chronic periodontitis, Local drug delivery,
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Atorvastatin (Active Comparator): 1.2% atorvastatin local drug delivery
  Interventions: Drug: 1.2% Atorvastatin local drug delivery
- Simvastatin (Sham Comparator): 1.2% simvastatin local drug delivery
  Interventions: Drug: 1.2% simvastatin local drug delivery
- Placebo (Placebo Comparator): Placebo local drug delivery
  Interventions: Drug: Placebo local drug delivery

INTERVENTIONS:
Drug: 1.2% Atorvastatin local drug delivery
  Arms: Atorvastatin
Drug: 1.2% simvastatin local drug delivery
  Arms: Simvastatin
Drug: Placebo local drug delivery
  Arms: Placebo

SUMMARY:
Background: Statins are the recently evolved agents that aid in periodontal regeneration and ultimately attaining periodontal health. Atorvastatin (ATV) and Simvastatin (SMV) are specific competitive inhibitors of 3-hydroxy-2-methyl-glutaryl coenzyme A reductase. The present study was designed to evaluate and compare the effectiveness of 1.2% ATV, and 1.2% SMV as an adjunct to scaling and root planing (SRP) in the treatment subjects with chronic periodontitis.

Methods: Ninety six subjects were categorized into three treatment groups: SRP plus 1.2% ATV, SRP plus 1.2% SMV and SRP plus placebo. Clinical parameters; full mouth plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD), and relative attachment level (RAL) were recorded at baseline before SRP and at 3, 6 and 9 months. Percentage radiographic defect depth reduction was evaluated using computer-aided software at baseline, 6 months and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe CP subjects with PD ≥ 5 mm or clinical attachment level (CAL) ≥ 4 mm and vertical bone loss ≥3 mm on intraoral periapical radiographs and no history of antibiotic or periodontal therapy in the preceding 6 months

Exclusion Criteria:

* Individuals with systemic diseases known to alter the course of periodontal disease and treatment outcome, known or suspected allergy to the SMV/ATV/statin group, those on systemic SMV/ATV/statin therapy, individuals with aggressive periodontitis, use of tobacco in any form, alcoholics, individuals with diabetes, immunocompromised individuals, and pregnant or lactating females

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in Radiographic intra-bony defect depth. | 9 months from baseline
  The primary outcome of the study was change in radiographic intra-bony defect depth from baseline to 9 months in all the groups. Intra-bony defect depth was measured on the radiograph by measuring the vertical distance from the crest of the alveolar bone to the base of the defect.

SECONDARY OUTCOMES:
Change in Probing depth. | 9 months from baseline
  Probing depth was measured from gingival margin to the base of pocket with a University of North Carolina no. 15 color-coded periodontal probe. change in probing depth was measured from baseline to 9 months.
Change in Relative attachment level | 9 months from baseline
  Relative attachment level was measured from a fixed point on the acrylic stent to the to the base of pocket. . A custom-made acrylic stent and a University of North Carolina no. 15 color-coded periodontal probe were used to standardize the measurement. Change was measured from baseline to 9 months.
Change in mSBI (gingival index) | 9 months from baseline
  modified sulcus bleeding index was measured at baseline and 9 months and the change in the values was taken as secondary outcome measure.
Change in plaque index | 9 months from baseline
  Sillness and loe plaque index was measured at baseline an 9 months and change in the values was taken as secondary outcome variable.

CONTACTS AND LOCATIONS:
Overall Officials: Avani R Pradeep, MDS, Principal Investigator — Professor